CLINICAL TRIAL: NCT04277897
Title: A Phase Ia Single-center,Randomized,Double-blind,Placebo-controled Study to Investigate the Safety, Tolerability, Pharmacokinetics of Single and Multiple Doses of Hepenofovir Fumarate Tablets in Healthy Volunteers.
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics of Single and Multiple Doses of Hepenofovir Fumarate Tablets in Healthy Volunteers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: XAXT-2019-001
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Drug SAD Cohorts (Experimental): Hepenofovir Fumarate Tablets Dose 1, Dose 2, Dose 3, Dose 4 and Dose 5 orally, once daily in one single administration.
  Interventions: Drug: Hepenofovir Fumarate Tablets Single Dose
- Placebo SAD Cohorts (Placebo Comparator): Matching placebo, orally, once daily in one single administration.
  Interventions: Drug: Placebo
- Drug MAD Group (Experimental): Hepenofovir Fumarate Tablets Dose 3 orally, once daily for 7 days.
  Interventions: Drug: Hepenofovir Fumarate Tablets Single Dose
- Placebo MAD Group (Placebo Comparator): Matching placebo, orally, once daily for 7 days.
  Interventions: Drug: Placebo
- Food-influnced Group (Experimental): Hepenofovir Fumarate Tablets Dose 4 orally, once daily in one single administration in fast condition,cross-over 7 days later in fed condition.
  Interventions: Drug: Hepenofovir Fumarate Tablets Dose4

INTERVENTIONS:
Drug: Hepenofovir Fumarate Tablets Single Dose — Oral Tablet; Subjects will receive either a single dose of Hepenofovir Fumarate Tablets on Day 1 only (SAD), once daily dosing of HTS starting on Day 1 through Day 7 (MAD).
  Arms: Drug MAD Group; Drug SAD Cohorts
Drug: Placebo — Placebo to match Hepenofovir Fumarate Tablets
  Arms: Placebo MAD Group; Placebo SAD Cohorts
Drug: Hepenofovir Fumarate Tablets Dose4 — Oral Tabet; Subjects will receive Hepenofovir Fumarate Tablets Dose4 on Day 1 in fast condition, then receive Hepenofovir Fumarate Tablets Dose4 on Day 8 in fed condition.
  Arms: Food-influnced Group

SUMMARY:
A Study to Investigate the Safety, Tolerability, Pharmacokinetics of Single and Multiple Doses of Hepenofovir Fumarate Tablets in Healthy Volunteers

DETAILED DESCRIPTION:
It's a single-center,randomized, double-blind, placebo-controlled study. It will assess the safety, tolerability, and pharmacokinetics of single and multiple orally administered doses of Hepenofovir Fumarate Tablets in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the nature of the study, comply with the protocol, and provide informed consent.
* Subjects willing to adhere to protocol requirements and to finish the study.
* Subjects were willing to use methods of contraception from the time of screen to 6 months post the last dose administration.
* Subjects aged between 18 and 55 years (both inclusive).
* Subject's weight within normal range according to normal values for Body Mass Index (19.00 to 26.00 kg/m2 (both inclusive)) ,with minimum of 50 kg weight for male, 45 kg weight for famale.
* Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within clinically acceptable normal range.

Exclusion Criteria:

* History or presence of significant smoking (more than 5 cigarettes/day prior to 3 months the first dose of the study drug).
* Hypersensitivity to different kinds of drugs and food.
* Presence of significant alcoholism or drug abuse.
* Volunteer who have donated blood or lose blood(>450mL)within past 90 days prior to the first dose of the study drug.
* Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 28 days prior to dosing of the study.
* Use of any prescribed medication or OTC medicinal products during the last 14 days prior to dosing of the study.
* Consumption of spcial food(including gragon fruit, mango, grapefruits) or strenuous excercise,or other factors which may effect the absorption,distribution,metabolism,excretion of drugs for within 2 weeks prior to dosing of the study.
* Any treatment which could bring about induction or inhibition of CYP3A4.
* Volunteer who have participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Difficulty in swallowing or other gastrointestinal disease or disorder.
* Presence of an abnormal electrocardiogram (ECG), which was clinically significant.
* Female subjects who were breast-feeding or had a positive pregnancy test at screening or at any time during the study.
* Subjects with abnormal health as determined by personal medical history, clinical examination and laboratory examinations,which was clinically significant.
* Subjects who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 6 Days in SAD Cohorts
Safety measured by adverse events | Up to 12 Days in MAD Group
Safety measured by adverse events | Up to 13 Days in Food-influence Group